CLINICAL TRIAL: NCT04397783
Title: Parastomal Hernia Prevention: Longitudinal Incision Versus Cruciate Incision in the Construction of an End Colostomy. LONG CROSS Trial
Brief Title: Longitudinal Incision Versus Cruciate Incision in the Construction of an End Colostomy
Acronym: LONGCROSS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Donostia (Other)
Responsible Party: Principal Investigator, Prof. Jose M Enríquez-Navascués, Professor, Hospital Donostia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ELO-HEP-2019-01
Record Dates: First submitted 2020-05-18; First posted 2020-05-21 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Colorectal Neoplasms; Parastomal Hernia; Colostomy Stoma
Keywords: end colostomy; colostomy; parastomal hernia; hernia prevention; prophylaxis; surgery; abdominal wall
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Masking Description: computer based aleatoric numbers
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cruciate incision (No Intervention): the classic cruciate incision in the colostomy construction
- longitudinal incision (Experimental): longitudinal incision with two proline sutures
  Interventions: Procedure: construction of an end colostomy

INTERVENTIONS:
Procedure: construction of an end colostomy — longitudinal incision in the construction of an end colostomy
  Other Names: colorectal surgery
  Arms: longitudinal incision

SUMMARY:
TITLE:

"Incidence of parastomal hernia: Randomized clinical trial comparing the longitudinal fascial incision (" Hepworth hitch ") vs. cruciate incision in the exteriorization of a end colostomy ".

DESIGN:

Randomized, open and parallel clinical trial so patients will be assigned to the cruciate incision group or longitudinal incision with a 1: 1 allocation ratio.

POPULATION:

Patients undergoing colorectal cancer surgery a definitive end colostomy.

OBJECTIVES:

The main objective is to compare the parastomal hernia rate diagnosed by imaging at 2 years after surgery.

Secondary objectives are:

1. Clinically relevant parastomal hernia rate by physical examination 2 years after surgery.
2. Incidence of postoperative complications related to the stoma (dehiscence, retraction, stenosis, necrosis, surgical revision, prolapse and special needs of care of the stoma in the immediate or late postoperative period); 3) Incidence of postoperative complications assessed according to the Comprehensive Complication Index (CCI) scale.

4) Ease / difficulty in the management of stomatherapy devices by patients using VAS (Visual Analogue Scale).

DESCRIPTION OF THE INTERVENTION:

An end colostomy without placement of a prophylactic mesh will be performed in all patients. In the group 1A, a longitudinal incision will be made in the anterior rectus fascia and in the posterior fascia, with two Prolene sutures at the ends of the incision of the anterior aponeurosis. In patients of group 1B, a cruciate incision will be made in the anterior rectus fascia, as well as in the posterior fascia.

DURATION OF THE STUDY:

The expected duration of the study is 3 years.

PATIENT FOLLOW UP TIME:

The planned follow-up time is 2 years.

EXPECTED RECRUITMENT TIME:

12 months.

DETAILED DESCRIPTION:
Parastomal hernia is one of the major complications after definitive terminal colostomy in patients with colorectal cancer, which is clinically relevant in up to 50% of the cases but can reach 78% of cases when radiologically identified. Although the majority of cases are asymptomatic, 26-30% of patients will require surgical intervention of the parastomal hernia for their symptoms, obstruction, incarceration, prolapse, leaks or aesthetic reasons.

Traditionally, the colostomy is made with a circular skin incision, dissection of the subcutaneous fat to the fascia and an incision of approximately 3 cm longitudinal and approximately 2 cm transversely. The anterior rectus muscle is loosened in the direction of the fibers and another cross incision is made in the posterior fascia to subsequently externalize the colon. The colostomy is fixed to the skin using mucocutaneous stitches of absorbable suture.

The hypothesis is that the longitudinal incision technique supplemented with Prolene stitches at the upper and lower ends of the incision acts as a "barrier" for the expansion of the hernia.

We designed a clinical trial to study the prevention of parastomal hernia with a simple modification such as making a vertical incision associated with four prolene stitches at the ends of incision, with minimal morbidity and an easy technique. The objective of the study is to analyze the postoperative parastomal hernia rate compared to the conventional technique (crossed incision).

JUSTIFICATION:

The longitudinal incision with prolene stitches at the ends of the incision is an easy and reproducible technique, with minimal morbidity. This technique is based on the theory that the hernia is a dilation of the hole that the surgeon has created. A vertical incision with two non-absorbable stitches at the ends would prevent the hole from dilating, since these act as a "barrier". This technique is related to a lower rate of parastomal hernias.

The objective of the study is to analyze if there are differences in the rate of parastomal hernias, clinically and radiologically measured without increasing postoperative morbidity.

POTENTIAL RISKS AND BENEFITS

Both techniques, the vertical incision and the crossed incision are approved techniques that are performed in a standardized way in most centers. There are no potential risks associated with the study intervention, beyond the intrinsic risks of the surgical intervention itself.

OBJECTIVES OF THE STUDY:

1. The main objective is to compare the rate of parastomal hernia diagnosed by image 2 years after surgery.
2. Secondary objectives are:

   * Clinically relevant parastomal hernia rate by physical examination 2 years after surgery.
   * Incidence of postoperative complications related to the stoma (dehiscence, retraction, stenosis, necrosis, surgical revision, prolapse and special needs for stoma care in the immediate or late postoperative period);
   * Incidence of postoperative complications assessed according to the Clavien-Dindo scale 10 and the Comprehensive Complication Index (CCI) 11.
   * Ease / difficulty for the handling of stoma therapy devices by patients using the Visual Analogue Scale (VAS)

   Clavien-Dindo Scale: The therapy used to correct a specific complication is the basis of this classification in order to rank a complication in an objective and reproducible manner.

   Grade I: any deviation from the normal postoperative course without the need for pharmacological treatment.

   Grade II: requiring pharmacological treatment with drugs other than such allowed for grade I complications. Blood transfusions and total parenteral nutrition are also included.

   Grade III: requiring surgical, endoscopic or radiological intervention. Grade IV: life-threatening complication requiring ICU management. Grade V: death of the patient.

   Comprehensive complication index (CCI): is based on the complication grading by Clavien-Dindo Classification and implements every occurred complication after an intervention. The overall morbidity is reflected on a scale from 0 (no complication) to 100 (death).

   Visual analogue scales (VAS) is psychometric measuring instrument designed to document the characteristics of disease-related symptom severity in individual patients and use this to achieve a rapid (statistically measurable and reproducible) classification of symptom severity and disease control, measuring from 0 (unhappy) 10 (very happy).

   STUDY OUTCOME MEASURES

   The following variables will be collected:

   • Demographic: sex, date of birth, weight, height, BMI, abdominal circumference, medical history (COPD, DM, respiratory failure, etc.), surgical history, date of tumor diagnosis, neoadjuvant treatment.
   * Preoperative evaluation: incisional hernia or previous hernias, previous abdominal surgeries, previous stoma.
   * Surgical treatment: date of surgical intervention, antibiotic prophylaxis, type of surgical approach, surgical team, mechanical bowel preparation, type of surgery (Hartmann intervention or abdominoperineal resection), descent of the splenic angle, stoma measurements, need for transfusion, duration of the intervention, bleeding, intraoperative complications.
   * Postoperative evolution: postoperative complications, date of diagnosis, reoperation, colostomy stenosis, colostomy prolapse, transfusion, hospital stay, postoperative mortality, and readmission.

   Evolution and follow-up: radiological or clinical parastomal hernia at one month, 12 months and 24 months.

   STUDY DESIGN

   • Randomized clinical trial, with a ratio of 1: 1, controlled, single-blind (the patient) of patients undergoing colorectal cancer who undergo a terminal colostomy without mesh.

   • The study population is patients hospitalized in participating centers with colorectal cancer, who underwent Hartmann's intervention, Miles' abdominoperineal amputation or Intersphincteric amputation, with definitive terminal colostomy.

   • Multicenter trial.

   • The expected recruitment period is 12 months. The follow-up time of the patients in the study is 24 months.

   • The approximate duration of the study is 3 years.

   Sample size calculation:

   According to published clinical trials and systematic reviews, up to 50% of patients with a terminal colostomy will develop a parastomal hernia. The estimated risk based on the publication by Manook et al, with the longitudinal incision of the fascia and Hepworth stitches is 10%. With the confidence level to 95% and a statistical power of 80% and having an expected loss ratio of 10% in each group, the sample size should be 21 in each group.

   Randomization process:

   Patients who meet the inclusion criteria for the study will be randomized using random number generating functions with the SPSS v.25 program in the longitudinal incision group or the crossed incision group. The randomization will be 1: 1 and will be stratified by the participating centers.

   The allocation will be concealed by means of sealed opaque envelopes. The envelope will be opened in the operating room at the beginning of the surgical intervention.

   Masking process:

   The patients do not know the intervention group to which they have been assigned. The surgeons and researchers know the group to which the patient has been assigned.

   DESCRIPTION OF THE STUDY INTERVENTION
   * General considerations in all patients included in the study:
   * Lithotomy position when doing the colostomy, regardless of whether it is subsequently modified in the prone position. Surgery by laparotomy or laparoscopy, performing Hartmann's Intervention or Abdominoperineal Amputation.
   * Balanced general anesthesia, with or without epidural catheter. Avoid volume overload and promote normothermia.
   * Usual positioning of the trocars (modifiable according to the surgeon's preferences). The extraction of the piece will be performed by a Minipfannenstiel, laparotomy or perineum, not through the colostomy incision.
   * The descent of the splenic angle must be total / partial / nule at the surgeon's discretion, but it must be stated in the notebook.
   * All patients participating in the study should undergo a colostomy in an area previously marked by a stomatherapist.
   * The colostomy is preferably externalized through the rectus abdominis muscle, but the externalization of the colostomy through the external oblique muscle is not an exclusion criterion, it must be stated in the notebook.
   * In the longitudinal incision group, the incision will be made on the aponeurosis of the anterior rectum of about 3 cm in length, without making any transverse incision. Depending on the diameter of the colon, two simple stitches of a 2/0 Prolene suture will be made at each end of the incision.
   * In the group of the cross incision, a longitudinal incision will be made on the aponeurosis of the anterior rectus or external oblique, about 3 cm long and another transverse incision, about 2 cm long, 1 cm on each side.
   * The length of the incision of the fascia must be recorded in the notebook.
   * The colostomy will be fixed to the skin with absorbable stitches, at the surgeon's discretion.
   * The fast track principles approved by different participating centers will be applied.

   STUDY CALENDAR (SCHEDULE)

   Colorectal cancer patients will be visited at outpatients. If the patient meets inclusion criteria, informed consent will be obtained in Outpatient Consultations, during colostomy marking or during admission prior to surgery.

   Preoperative study period:
   * PRELIMINARY PHASE: Preparation of data collection form.
   * RECRUITMENT PHASE (12 months):

   Visit -1 Colorectal cancer patients who are going to have a terminal colostomy are visited in the outpatient clinic. If the patient meets inclusion criteria, the clinical trial will be explained and the informed consent will be signed. The stomatherapist marks the stoma site prior to surgery.

   Visit 0 It will be confirmed that the patient has signed the informed consent. It will be verified that the patient meets the inclusion criteria. Baseline data and confounding factors described in the variables will be obtained.

   In the operating room, the randomization envelope will be opened and the surgical technique will be performed.

   Visit +1 Postoperative variables will be collected: stoma status, postoperative complications, reoperations, transfusions, hospital stay, postoperative mortality, and readmission.

   • FOLLOW-UP PHASE (24 months): Obtaining the data and variables will be obtained on visits to the first month, 12th and 24th month. A clinical and radiological examination will be performed at each consultation. The patient must complete the corresponding questionnaires. BMI and abdominal circumference will be measured in control visits.

   • PUBLICATION PHASE (6 months): Preparation of the article for the publication of the results: 6 months after the process of data collection and statistical analysis finished.

   •DISTRIBUTION OF TASKS: The patients included in the study will be randomized. One of the main researchers will be responsible for the study design and analysis. The research group as a whole is responsible for preparing the publication of the results obtained.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing surgery for colorectal cancer undergoing definitive end colostomy.
* Age ≥ 18 years and <85 years.
* Any type of tumor, any T, N, M0.
* Consent signed by the patient and by the researcher.

Exclusion Criteria:

* no colostomy, not end stoma.
* Inflammatory bowel disease with anatomopathological confirmation.
* Patients with previous incisional hernias or carriers of meshes except inguinal hernioplasties.
* Patients with previous stoma.
* Inability to read or understand any of the languages of informed consent.
* Emergency surgery.
* Psychiatric diseases, addictions or any disorder that prevents the compression of informed consent.
* Extraction of the piece by colostomy hole.
* Colostomies not previously marked by specialized stomatherapist.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2019-04-15 (Actual); Primary Completion 2019-10-15 (Actual); Study Completion 2022-04-15 (Estimated)

PRIMARY OUTCOMES:
parastomal hernia rate by imaging | 2 years
  parastomal hernia by CT

SECONDARY OUTCOMES:
Clinically relevant parastomal hernia rate | 2 years after surgery
  by physical examination
Incidence of postoperative complications related to the stoma (dehiscence, retraction, stenosis, necrosis, surgical revision, prolapse and special needs | 2 years
  Physical examination
Ease / difficulty in the management of stomatherapy devices | 2 years
  using VAS scale (Visual Analogue Scale). Visual analogue scales (VAS) is psychometric measuring instrument designed to document the characteristics of disease-related symptom severity in individual patients and use this to achieve a rapid (statistically measurable and reproducible) classification of symptom severity and disease control, measuring from 0 (unhappy) 10 (very happy).

CONTACTS AND LOCATIONS:
Locations (1):
- Jose Maria Enriquez Navascues, Donostia / San Sebastian, Spain

IPD SHARING:
Plan to Share IPD: Undecided